CLINICAL TRIAL: NCT02745938
Title: GDF-15 as a Biomarker for Mitochondrial Disease
Acronym: GDF-15
Status: Completed | Type: Observational
Sponsor: Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Nanna Scharff Nielsen, Student researcher, Rigshospitalet, Denmark
Other Study IDs: H-16023953
Record Dates: First submitted 2016-04-12; First posted 2016-04-20 (Estimated); Last update posted 2017-08-17 (Actual); Status verified 2017-08

CONDITIONS: Mitochondrial Disease; Metabolic Myopathy; Muscular Dystrophy
Keywords: Exercise test; GDF-15; Growth and Differentiation Factor 15
MeSH Terms: conditions — Mitochondrial Diseases; Muscular Dystrophies

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Blood samples
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (4):
- Mitochondrial disease: Patients with mitochondrial disease, investigated by blood samples and exercise test.
- Metabolic myopathy: Patients with metabolic myopathy, investigated by blood samples and exercise test.
- Muscular dystrophy: Patients with muscular dystrophy, investigated by blood samples and exercise test.
- Healthy controls: Healthy controls, investigated by blood samples and exercise test.

SUMMARY:
Mitochondrial disorders are a group of inherited disorders causing malfunctional mitochondria. Mitochondria are found in every cell of the body, and the disorders therefore give symptoms from every tissue, especially those with high energy needs as the brain, heart and muscles. The symptoms are often unspecific in terms of muscle weakness and fatigue, which delays the first contact to the doctor and further delays the diagnosis.

The aim of this study is to investigate if it is possible to use GDF-15 (Growth and Differentiation Factor 15) as a biomarker for mitochondrial disease and compare the results with that of healthy controls, metabolic myopathies and muscular dystrophies. The concentration relative to exercise will further be investigated.

DETAILED DESCRIPTION:
BACKGROUND

Energy insufficiency:

Mitochondrial and metabolic myopathies are inherited diseases compromising cellular energy metabolism, which especially affects skeletal muscle because of its high energy needs. Chemical energy is stored in the body as adenosine triphosphate (ATP), which is derived from different sources including breakdown of carbohydrates, lipids and purine nucleotides. In the respiratory chain in the inner mitochondrial membrane, ATP is released through oxidative phosphorylation.

Any genetic disorder affecting any step in the production of energy, from storage and breakdown of glycogen and lipids to transport and conversion of substrates, can manifest as energy insufficiency in the affected tissues.

Mutations in genes encoding enzymes of the lipid or carbohydrate metabolism result in metabolic myopathies and mutations in the enzyme complexes of the respiratory chain result in mitochondrial disorders.

Mitochondrial disorders:

Mitochondrial disorders are caused by mutations in either mitochondrial DNA (mtDNA) or nuclear DNA (nDNA) which lead to impaired function of the respiratory chain and reduced energy generation. The disorders derived from mtDNA mutations are maternally inherited, while the nDNA mutations are autosomal recessively or dominantly inherited.

Mitochondrial disorders present with a wide range of symptoms and syndromes depending on the mutation and mutation load in tissues. Symptoms usually arise from the brain, nerves, skeletal and cardiac muscle, as these tissues have a high energy demand. The patients may suffer from muscle weakness, exercise intolerance, impaired balance and coordination, seizures, learning deficits, impaired vision, hearing loss and heart defects. Age at disease onset varies and the disease can debut throughout life.

The prevalence is in general 6.2/100.000 births.

Metabolic myopathies:

Metabolic myopathies are either inherited autosomal recessively, dominantly, X-linked or occur spontaneously. Metabolic myopathies can be caused by defective enzymes of the lipid metabolism (Fatty Acid Oxidation Disorders), and glycogen and glucose metabolism (Glycogenoses) with common features of compromised energy generation in the affected tissues, especially in muscle.

Symptoms vary, but patients can suffer from exercise intolerance, muscle contractures, progressive muscle weakness and heart- and respiratory failure. If the symptoms start in childhood, the disease is often more severe and may present with acute metabolic decompensation, hypoketotic hypoglycemia, encephalopathy and risk of coma and death.

The prevalence and incidence are uncertain, since there might be many patients who have not been diagnosed. With an increased awareness and newborn screening programs, more patients are now being diagnosed and survive metabolic decompensation.

Growth Differentiation Factor 15 as a diagnostic tool:

Since the symptoms of mitochondrial disorders and metabolic myopathies are very unspecific, they can easily be mistaken for i.e. cardiopulmonary disease and diagnosis can be difficult. Therefore, it would be useful to have a biomarker that could easily distinguish both disorders from others. A recent study showed that Growth Differentiation Factor 15 (GDF-15) was significantly elevated in blood from patients affected by mitochondrial disorders as compared to healthy individuals, but it is unknown whether this increase is specific for mitochondrial disease. Thus it is unknown how GDF-15 levels are in patients with other muscle disease, including metabolic myopathies in which an energy deficiency, as in mitochondrial diseases, is also present. GDF-15 belongs to the transforming growth factor beta super family of growth factors that regulates inflammation and apoptosis in injured tissue. It is not known why GDF-15 is elevated, but it has been suggested that the oxidative stress, which is a part of the pathophysiology in mitochondrial disorders, increases GDF-15 through activation of P53. Oxidative stress also plays a role in the pathophysiology of some metabolic myopathies [8], and GDF-15 may therefore be elevated in these patients too. To make sure that the GDF-15 is not elevated due to muscle involvement, it will also be measured in a subgroup of muscular dystrophies.

AIM

In this study, we wish to further investigate:

1. if measurement of GDF-15 can be used as a biomarker for mitochondrial myopathy and distinguish these patients from healthy persons.
2. if elevated GDF-15 is also a sign of either metabolic myopathy or muscle dystrophy and not exclusively detects mitochondrial disease.
3. if the GDF-15 concentration in these mitochondrial and metabolic myopathy varies when metabolic demand is increased with exercise.
4. if the GDF-15 concentration correlates with oxidative capacity (VO2max) in patients with mitochondrial myopathy.

We will investigate the concentration of GDF-15 in blood samples in patients affected by mitochondrial disorders and compare it to the concentrations in patients affected by metabolic myopathies, muscular dystrophies and to a group of healthy controls. If there is a significant difference, GDF-15 may be a sensitive biomarker for mitochondrial disorders. We will further investigate the maximal oxidative capacity and the maximal workload capacity to study if and how this relates to the concentration of GDF-15.

METHODS:

30 subjects with mitochondrial disorders, 25 with metabolic myopathy, 25 with muscular dystrophy and 25 healthy controls will be recruited. A blood sample will be taken, and GDF-15 and other muscle markers will be measured. 10-15 subjects with mitochondrial disorders, 10-15 with metabolic myopathy and 10-15 healthy individuals will further be investigated with an exercise test, and blood samples will be taken afterwards.

ELIGIBILITY:
Criteria for subjects with mitochondrial disease, metabolic myopathy or muscle dystrophy:

Inclusion Criteria:

* Verified mitochondrial disease, metabolic myopathy or muscular dystrophy.

Exclusion Criteria:

* Other muscle disorders.
* Heart failure or significantly reduced kidney or lung function.
* Contraindications for exercise test, e.g. serious heart and lung disease. The investigator will decide whether or not it is possible for the subject to participate (Only for the subjects doing an exercise test.).

Criteria for healthy individuals:

Inclusion Criteria:

None (except age > 15 years).

Exclusion Criteria:

* Any muscle disorder
* Heart failure
* Contraindications for exercise test, e.g. serious heart and lung disease. The investigator will decide whether or not it is possible for the subject to participate (Only when participating in the exercise test).

Min Age: 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Four groups are studied:
  1. Patients with mitochondrial disease.
  2. Patients with metabolic myopathy.
  3. Patients with muscular dystrophy.
  4. Healthy controls.
Sampling Method: Non-Probability Sample
Enrollment: 97 (Actual)
Dates: Start 2016-06; Primary Completion 2017-08 (Actual); Study Completion 2017-08 (Actual)

PRIMARY OUTCOMES:
GDF-15 concentration in plasma sample at rest. | One blood sample per subject will be analysed. It takes 5 minutes.
  The blood sample will be analysed with a Luminex analyser to determine the concentration of GDF-15.

SECONDARY OUTCOMES:
GDF-15 concentration in plasma after exercise | The exercise test takes half an hour. Blood samples will be taken 1, 2, 3, 24 and 48 hours after the exercise test.
  The subjects perform an incremental exercise test until exhaustion on a cycle ergometer. The concentration of GDF-15 is measured afterwards with a Luminex analyser.
Other biomarkers of energy metabolism disorders at rest and after exercise test. | If the blood samples are only taken at rest, the test takes 5 minutes. If an exercise test is done, it takes 48 hours.
  Lactate is a muscle marker, that is measured in this study.
Other biomarkers of energy metabolism disorders at rest and after exercise test. | If the blood samples are only taken at rest, the test takes 5 minutes. If an exercise test is done, it takes 48 hours.
  Pyruvate is a muscle marker, that is measured in this study.
Other biomarkers of energy metabolism disorders at rest and after exercise test. | If the blood samples are only taken at rest, the test takes 5 minutes. If an exercise test is done, it takes 48 hours.
  Creatin kinase is a muscle marker, that is measured in this study.
Other biomarkers of energy metabolism disorders at rest and after exercise test. | If the blood samples are only taken at rest, the test takes 5 minutes. If an exercise test is done, it takes 48 hours.
  FGF-21 (Fibroblast Growth Factor 21) is a muscle marker that is measured in this study.
Maximal oxidative capacity (VO2max) | The test takes half an hour per subject.
  During the exercise test, the subjects will breath through a mask, that is connected to a machine. The machine is able to calculate the VO2max.
Maximal workload capacity (Wmax) | The test takes half an hour per subject.
  The Wmax will be calculated during the exercise test.

CONTACTS AND LOCATIONS:
Overall Officials: Nanna S. Nielsen, B.Sc., Principal Investigator — Copenhagen Neuromuscular Center
Locations (1):
- Rigshospitalet, Copenhagen, Copenhagen East., Denmark

IPD SHARING:
Plan to Share IPD: No
No plan

REFERENCES:
- [Background] Sharp LJ, Haller RG. Metabolic and mitochondrial myopathies. Neurol Clin. 2014 Aug;32(3):777-99, ix. doi: 10.1016/j.ncl.2014.05.001. PMID 25037090
- [Background] Lightowlers RN, Taylor RW, Turnbull DM. Mutations causing mitochondrial disease: What is new and what challenges remain? Science. 2015 Sep 25;349(6255):1494-9. doi: 10.1126/science.aac7516. Epub 2015 Sep 24. PMID 26404827
- [Background] Yatsuga S, Fujita Y, Ishii A, Fukumoto Y, Arahata H, Kakuma T, Kojima T, Ito M, Tanaka M, Saiki R, Koga Y. Growth differentiation factor 15 as a useful biomarker for mitochondrial disorders. Ann Neurol. 2015 Nov;78(5):814-23. doi: 10.1002/ana.24506. Epub 2015 Oct 14. PMID 26463265
- [Background] Kalko SG, Paco S, Jou C, Rodriguez MA, Meznaric M, Rogac M, Jekovec-Vrhovsek M, Sciacco M, Moggio M, Fagiolari G, De Paepe B, De Meirleir L, Ferrer I, Roig-Quilis M, Munell F, Montoya J, Lopez-Gallardo E, Ruiz-Pesini E, Artuch R, Montero R, Torner F, Nascimento A, Ortez C, Colomer J, Jimenez-Mallebrera C. Transcriptomic profiling of TK2 deficient human skeletal muscle suggests a role for the p53 signalling pathway and identifies growth and differentiation factor-15 as a potential novel biomarker for mitochondrial myopathies. BMC Genomics. 2014 Feb 1;15:91. doi: 10.1186/1471-2164-15-91. PMID 24484525
- [Background] Kitaoka Y, Ogborn DI, Nilsson MI, Mocellin NJ, MacNeil LG, Tarnopolsky MA. Oxidative stress and Nrf2 signaling in McArdle disease. Mol Genet Metab. 2013 Nov;110(3):297-302. doi: 10.1016/j.ymgme.2013.06.022. Epub 2013 Jul 6. PMID 23906480
- [Background] Suomalainen A, Elo JM, Pietilainen KH, Hakonen AH, Sevastianova K, Korpela M, Isohanni P, Marjavaara SK, Tyni T, Kiuru-Enari S, Pihko H, Darin N, Ounap K, Kluijtmans LA, Paetau A, Buzkova J, Bindoff LA, Annunen-Rasila J, Uusimaa J, Rissanen A, Yki-Jarvinen H, Hirano M, Tulinius M, Smeitink J, Tyynismaa H. FGF-21 as a biomarker for muscle-manifesting mitochondrial respiratory chain deficiencies: a diagnostic study. Lancet Neurol. 2011 Sep;10(9):806-18. doi: 10.1016/S1474-4422(11)70155-7. Epub 2011 Aug 3. PMID 21820356